CLINICAL TRIAL: NCT04324060
Title: A Randomized Trial of Recombinant Human Thrombopoietin Versus Placebo for Low/Intermediate-1 Risk Myelodysplastic Syndromes With Thrombocytopenia
Brief Title: A Randomized Trial of rhTPO Versus Placebo for Low/Intermediate-1 Risk MDS With Thrombocytopenia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TPO
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Low/Intermediate Risk-1 MDS
MeSH Terms: interventions — Danazol; Thrombopoietin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPO treatment group (Active Comparator): Danazol 0.2g tid po+rhTPO (recombinant human thrombopoietin injection) 300U/kg/d×14d si every month (stop when PLT≥100×10e9/L or increased more than 50×10e9/L), total course 6 months
  Interventions: Drug: Danazol + rhTPO (recombinant human thrombopoietin injection)
- control (Placebo Comparator): Danazol 0.2g tid po+ control (sodium chloride)×14d si every month, total course 6 months
  Interventions: Drug: Danazol + sodium chloride

INTERVENTIONS:
Drug: Danazol + rhTPO (recombinant human thrombopoietin injection) — subcutaneous injection, 300U/kg/d×14d every month，stop if the PLT≥100×10e9/L or increased >50×10e9/L, total course is 6 months
  Arms: TPO treatment group
Drug: Danazol + sodium chloride — Danazol 0.2g tid po+ control (sodium chloride)
  Arms: control

SUMMARY:
Myelodysplastic syndrome (MDS) is a kind of clonal myeloid tumor. The major manifestation is decrease of tri-lineages of blood due to ineffective and abnormal hematopoiesis, some of which can progress to acute myeloid leukemia. According to the international prognosis scoring system (IPSS) of MDS, about 10% low/intermediate risk-1 MDS patients have severe thrombocytopenia (PLT < 30 × 109/ L). These patients have both decreased platelet count and platelet dysfunction, resulting in a high risk of bleeding. In the new prognostic score, such as IPSS-r, the degree of thrombocytopenia is regarded as a poor prognostic factor. Platelet transfusion is mainly used in the treatment of this kind of patients. The indications of transfusion include bleeding events or severe platelet count reduction (< 10 × 109 / L). However, platelet transfusion can only lead to short-term platelet elevation, while repeated transfusion increases the possibility of infection and ineffective platelet transfusion. TPO is a newly discovered hematopoietic promoting factor, which can specifically bind to the TPO receptor on the cell and participate in the regulation of proliferation, differentiation, maturation and division of megakaryocyte to form functional platelet. The efficacy and safety of the TPO receptor agonists eltrombopag and romiplostim in the treatment of thrombocytopenia in low/intermediate risk-1 MDS patients have been successfully confirmed in foreign studies. Recombinant human thrombopoietin (rhTPO) is also a kind of a TPO receptor agonists which is highly specific platelet stimulating factor. At present, there is no large report on the application of rhTPO in such patients. The purpose of this study is to explore the short-term and long-term therapeutic effect and safety of rhTPO on low/intermediate risk-1 MDS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed MDS, IPSS low / intermediate risk-1
2. In the 4 weeks before inclusion, the average value of platelets was ≤ 30 × 10e9 / L, or < 50 × 10e9 / L with bleeding events
3. Patients with EPO due to anemia and G-CSF due to severe neutropenia can be included, and the dosage will not change during trial
4. Baseline liver and kidney function: ALT / ASL within 3 times normal upper limit, TBIL within 2 times normal upper limit, and creatinine within 2 times normal upper limit
5. ECOG 0-2 points
6. Able to sign informed consent

Exclusion Criteria:

1. Pregnant or lactating
2. IPSS intermediate risk-2 / high risk MDS
3. More than 5% of myeloblasts in bone marrow
4. Myelofibrosis
5. Previous transplantation or ATG treatment within 6 months
6. Previous use of IL-11, TPO or other TPO receptor agonists
7. Active infection or tumor
8. Thromboembolic or hemorrhagic disease
9. Serious heart disease, including unstable angina, congestive heart failure, arrhythmia, 1-year history of myocardial infarction
10. Intracranial hemorrhage within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 1 year
  overall response rate of platelet
rate of side effects | 1 year
  rate of all kinds of side effects

SECONDARY OUTCOMES:
WHO bleeding score | 1 year
  to evaluate frequency and severity of bleeding
change of platelet transfusion | 1 year
  the frequency and amount of platelet transfusion
onset time for overall response | through study completion, an average of 1 year
  onset time for complete and partial response
duration of overall response | through study completion, an average of 1 year
  during time for complete and partial response
incidence of TPO antibody | 1 year
  rate of presence of TPO antibody
life quality for MDS patients | 1 year
  life quality for MDS patients by QoL-E questionaire
the increased number of myeloblasts in bone marrow and peripheral blood | 1 year
  the increased number of myeloblasts in bone marrow and peripheral blood
incidence of progression to high-risk MDS or leukemia | 1 year
  incidence of progression to high-risk MDS or leukemia

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
protocol, consent form, clinical data would be available by personal contact
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 10 years
Access Criteria: personal contact including emails

REFERENCES:
- [Derived] Yang Y, Tang Z, Ji J, Yang C, Chen M, Han B. Recombinant Human Thrombopoietin Accelerates the Recovery of Platelet in Patients With Lower-Risk Myelodysplastic Syndrome: A Proof-of-Concept Study. Front Oncol. 2021 Oct 28;11:721764. doi: 10.3389/fonc.2021.721764. eCollection 2021. PMID 34778037